CLINICAL TRIAL: NCT05131750
Title: A Prospective Study of Residual Inflammatory Risk and the Impact on Clinical Outcomes in Patients Undergoing Percutaneous Coronary Interventions
Brief Title: RIR and the Impact on Clinical Outcomes in Patients Undergoing PCI
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiang Cheng, Head of department of cardiology, Wuhan Union Hospital, China, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Other Study IDs: RIR-PCI
Record Dates: First submitted 2021-05-03; First posted 2021-11-23 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: hsCRP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coronary heart disease (CAD) is caused by myocardial ischemia, hypoxia or necrosis due to coronary artery stenosis, spasm or obstruction. Although standard drug therapy can greatly improve the prognosis of patients with CAD after percutaneous coronary interventions (PCI), these patients are still at high risk of major adverse cardiovascular events (MACE).

At present, the concept of residual inflammation risk (RIR) has aroused widespread concern. RIR is an important independent risk in patients with CAD. Foreign studies indicate that hsCRP ≥ 2mg / L is the definition standard of RIR in CAD. In China, there is no defined value of RIR for patients undergoing PCI, and the incidence of RIR has not been investigated clearly. At the same time, the impact of dynamic changes of hsCRP on MACE in PCI population needs to be further explored. Therefore, in this study, we plan to recruit patients undergoing PCI, and observe the impact of RIR by serial hsCRP measurements on the prognosis of these patients followed up for 5 years.

DETAILED DESCRIPTION:
Serial hsCRP measurements with ≥ 4 weeks between both measurements are defined in this analysis. Time-to-event is measured from first hsCRP measurement.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who understand and sign the informed consent form voluntarily;
2. Age ≥ 18 years old and ≤ 80 years old, regardless of sex;
3. The hospitalized patients with coronary heart disease undergoing PCI;
4. Complete all planned PCI during hospitalization

Exclusion Criteria:

1. Patients do not receive standardized treatment according to guidelines after being diagnosed with coronary heart disease;
2. Uncontrolled infectious diseases during the screening period;
3. In the screening stage, patients with immune diseases or immune-related diseases such as systemic lupus erythematosus, asthma, inflammatory bowel disease, gout, malignant tumor and so on;
4. Long-term use of non-steroidal anti-inflammatory drugs, hormones, immunomodulatory and chemotherapeutic drugs during the study period;
5. Surgical or interventional treatment was performed within 3 months before the screening period;
6. Pregnant women, lactating women or women of childbearing age who do not use effective contraceptives;
7. Participated in other clinical trials within 3 months before the screening period;
8. The researchers determined that other conditions in which the patient was not suitable to participate in the clinical trial.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with coronary heart disease completed all planned PCI during hospitalization
Sampling Method: Probability Sample
Enrollment: 1408 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACEs) | 60 months
  Composite endpoint of all-cause death, nonfatal myocardial infarction, nonfatal stroke, and revascularization due to ischemia

SECONDARY OUTCOMES:
All-cause death | 60 months
  Death due to any cause
Cardiovascular death | 60 months
  Death due to cardiovascular cause
Nonfatal myocardial infarction | 60 months
  According to the fourth edition of the General Definition of Myocardial Infarction
Revascularization due to ischemia | 60 months
  Ischemia driven revascularization, including repeated PCI or CABG due to recurrent or persistent ischemic symptoms
In-stent thrombosis | 60 months
  In-stent thrombosis is determined based on the degree of certainty and the time after PCI
Nonfatal stroke | 60 months
  Acute neurological deficits caused by pathological basis of cerebral infarction, cerebral hemorrhage, subarachnoid hemorrhage, and cerebral venous sinus thrombosis affecting brain tissue
Bleeding | 60 months
  According to the report from the Bleeding Academic Research Consortium

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Result] Ridker PM, Everett BM, Thuren T, MacFadyen JG, Chang WH, Ballantyne C, Fonseca F, Nicolau J, Koenig W, Anker SD, Kastelein JJP, Cornel JH, Pais P, Pella D, Genest J, Cifkova R, Lorenzatti A, Forster T, Kobalava Z, Vida-Simiti L, Flather M, Shimokawa H, Ogawa H, Dellborg M, Rossi PRF, Troquay RPT, Libby P, Glynn RJ; CANTOS Trial Group. Antiinflammatory Therapy with Canakinumab for Atherosclerotic Disease. N Engl J Med. 2017 Sep 21;377(12):1119-1131. doi: 10.1056/NEJMoa1707914. Epub 2017 Aug 27. PMID 28845751
- [Result] Kalkman DN, Aquino M, Claessen BE, Baber U, Guedeney P, Sorrentino S, Vogel B, de Winter RJ, Sweeny J, Kovacic JC, Shah S, Vijay P, Barman N, Kini A, Sharma S, Dangas GD, Mehran R. Residual inflammatory risk and the impact on clinical outcomes in patients after percutaneous coronary interventions. Eur Heart J. 2018 Dec 7;39(46):4101-4108. doi: 10.1093/eurheartj/ehy633. PMID 30358832
- [Result] Ridker PM. Residual inflammatory risk: addressing the obverse side of the atherosclerosis prevention coin. Eur Heart J. 2016 Jun 7;37(22):1720-2. doi: 10.1093/eurheartj/ehw024. Epub 2016 Feb 22. No abstract available. PMID 26908943